CLINICAL TRIAL: NCT05342922
Title: Comparison of Ultrasound and Anatomical Land-mark Method in Spinal Anesthesia for Elective Cesarean Section in Obese Parturients With BMI ≥ 40 kg/m2. A Randomized Controlled Trial
Brief Title: The Ultrasound Guided Versus Land-mark Location Method for Performing Spinal Anesthesia in Obese Parturients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karaman Training and Research Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-2022/02
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2022-04

CONDITIONS: Morbid Obesity
Keywords: Spinal Anesthesia; Cesarean Delivery; Ultrasound
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Allocation: Randomized Intervention Model: Parallel Assignment
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple (Participant,Investigator, Outcomes Assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound group (Active Comparator): Ultrasound assited technique will be used for spinal anesthesia performance.
  Interventions: Procedure: Ultrasound group
- Landmark group (Experimental): Land-mark assisted technique will be used for spinal anesthesia performance.
  Interventions: Procedure: Landmark group

INTERVENTIONS:
Procedure: Ultrasound group — In the operating room, all of the patients will receive standard monitoring. Scans will be made in logiditunal parasagittal and transverse midline views with ultrasound. Needle entry sites in the L2-L3 and L3-L4 intervals will be determined as the intersection of the longiditunal and transverse lines.
  When the spinal puncture operator is outside the room, Needle entry sites were marked for both groups.After skin marking, the pregnant woman will be asked to remain still and a subarachnoid puncture will be performed immediately. Spinal anesthesia will be administered with injection of intrathecal bupivacaine.
  Arms: Ultrasound group
Procedure: Landmark group — In the Landmark group, the injection site will be determined using the traditional method of palpating the posterior superior iliac spine.When the spinal puncture operator is outside the room, Needle entry sites were marked for both groups.After skin marking, the pregnant woman will be asked to remain still and a subarachnoid puncture will be performed immediately. Spinal anesthesia will be administered with injection of intrathecal bupivacaine.
  Arms: Landmark group

SUMMARY:
This study will be investigated whether an ultrasound-assisted technique is better than a classical land-mark technique to facilitate spinal anesthesia in the lateral position in morbidly obese pregnant women with BMI ≥ 40 who will undergo elective cesarean section.

The primary objective in this study is the rate of successful dural puncture at the first attempt. It was assumed that ultrasound could facilitate neuraxial blockade in grade 3 morbidly obese pregnant women according to the Who classification, whose topographic anatomy is difficult.

DETAILED DESCRIPTION:
Spinal anesthesia is the most commonly used anesthesia method for elective cesarean deliveries. Anesthesiologists may have difficulties in determining the poorly palpable surface landmarks in morbidly obese pregnant women.

Manual palpation technique, which is preferred in neuraxial anesthesia, may be difficult in obese pregnant women due to the difficulty in identifying bone landmarks. Neuraxial ultrasound examination before spinal anesthesia may help spinal anesthesia performance and decrease number of attempts in obese parturients.

This study will be conducted as a single-center, prospective, randomized, double-blinded trial in a university hospital. Patients scheduled for elective cesarean will be screened for enrollment in the study. Patient, the anesthetist administering spinal anesthesia and evaluating the data were blind to the distribution of patient groups.Ultrasonographic examinations were performed by a single investigator trained in this technique who performed more than 150 ultrasound-guided neuraxial blocks.

ELIGIBILITY:
Inclusion Criteria:

* Parturient who will receive selective cesarean delivery under spinal anesthesia
* ASA 2-3 scheduled for elective sections
* BMI≥40 kg/m2
* normal singleton pregnancy
* ≥37 weeks of gestation

Exclusion Criteria:

* Multiple gestations
* Emergency C-section
* exist contraindications of spinal anesthesia
* Local anesthetics allergy
* BMI<40 kg/m2
* history of lumbar spinal diseases and lumbar surgery
* Parturient refusal

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study only includes pregnant patients who will deliver by elective cesarean section.
Enrollment: 80 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-01-23 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
The success rate of first puncture | 30 minute
  Success on a single-puncture attempt will be defined as reaching the subarachnoid space on the first insertion of the needle.

SECONDARY OUTCOMES:
Number of skin punctures | 30 minute
  Skin puncture is defined as any separate skin puncture attempt.
Number of needle pass | 30 minute
  Needle pass is defined as skin puncture plus number of redirection attempts
The procedure duration time | 30 minute
  The duration from initiation of location marking by palpation or ultrasound to obtaining free cerebrospinal fluid flow
Time interval to determine needle insertion site | 30 minute
  Time interval between the operator touches the parturient and the completion of the needle insertion point marking
Time taken for spinal injection | 30 minute
  The time interval between the needle insertion to visualization of cerebrospinal spinal fluid in the spinal needle.
Number of puncture levels | 30 minute
  Move to a second lumbar space after 3 needle insertion attempts
Patient satisfaction The procedure duration | 30 minute
  Patients rated their satisfaction as very satisfied, satisfied, or dissatisfied immediately after the procedure.
incidence of complications during puncture | 30 minute
  Incidence of radicular pain, paresthesia, and blood during spinal needle injection
incidence of postoperative headache | 72 hour
  12-72 hours following spinal anesthesia due to CSF leakage
Incidence of hypotension | 2 hour
  A systolic arterial pressure decrease of more than 25% from baseline or less than 90 mmHg
Failure rate of spinal anesthesia | 120 minute
  Number of parturients who need additional analgesic drug or conversion to general anesthesia
dermatome level of sensory block [ Time Frame: 10 minutes after spinal anesthetic injection ] | 20 minute
  thoracic dermatome level of sensory block assessed by pinprick test

CONTACTS AND LOCATIONS:
Overall Officials: Betul Basaran, MD,DESA, Study Director — Karaman Training and Research Hospital
Locations (1):
- Karaman Training and Research Hospital, Karaman, Turkey (Türkiye)